CLINICAL TRIAL: NCT00396409
Title: A Randomized, 20 Week, Double-blind, Placebo-controlled, Parallel-group, Multiple-dose, Multicenter Study to Assess the Efficacy and Safety of Omalizumab in Combination With Depigoid, Versus Depigoid Only, in Adult and Adolescent Patients With Seasonal Allergic Asthma and Comorbid Seasonal Allergic Rhinoconjunctivitis - Open-label Depigoid Monotherapy Extension Periods 2007 and 2008-
Brief Title: Efficacy/ Safety of Omalizumab in Patients With Seasonal Allergic Asthma and Seasonal Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIGE025ADE03
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Depigold+Omalizumab (Experimental): Xolair® (Omalizumab, double-blind core study period only), Depigoid® (grass/rye pollen 50/50)
  Interventions: Drug: Depigoid; Drug: Omalizumab
- Depigoid+Placebo (Experimental): Depigoid® (grass/rye pollen 50/50) + Placebo
  Interventions: Drug: Depigoid; Drug: Placebo

INTERVENTIONS:
Drug: Depigoid — Administered in 4-week intervals using 0.5 ml of vial 2 (1000 DPP/mL)
Drug: Omalizumab — anti-IgE (Omalizumab) given during the 2006 core study
  Other Names: Xolair
  Arms: Depigold+Omalizumab
Drug: Placebo — Placebo given during the 2006 core study
  Arms: Depigoid+Placebo

SUMMARY:
Efficacy/ safety for the combination of anti-IgE (Omalizumab) and specific immunotherapy (Depigoid) in patients with not adequately controlled seasonal allergic asthma and comorbid seasonal allergic rhinoconjunctivitis.

DETAILED DESCRIPTION:
This was an open-label extension period of the previously randomized, multicenter, double-blind, placebo-controlled, parallel-group trial to demonstrate the benefit of pre- and co-seasonal combination therapy with anti-IgE (omalizumab) and specific immunotherapy (Depigoid) in patients with seasonal allergic asthma and co-morbid seasonal allergic rhinoconjunctivitis. During the open-label period, all patients received Depigoid monotherapy for two follow-up seasons every 4 weeks, 26 injections in total. The extension period was performed to evaluate the influence of omalizumab on the follow-up treatment with Depigoid in seasonal asthma.

This study was a follow-up to the core IGE025ADE03 study, in which patients received omalizumab treatment. In this follow-up study, no patient received omalizumab.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any race who are 12-45 years of age with a body weight ≥ 20 kg and ≤ 150 kg and with a total serum IgE level ≥ 30 to ≤ 700 IU/ml (suitable weight for dosing)
* Patients with the diagnosis of not adequately controlled seasonal grass pollen (and/or rye pollen) and allergic asthma with concomitant seasonal allergic rhinoconjunctivitis within > 2 previous seasons
* patients with a positive RAST (>CAP2) result for grass pollen (and/or rye pollen) specific IgE at screening (Visit 1 (V1) or within the previous 12 months.
* Patients with FEV1 > 80% of the predicted normal value for the patient at screening [V1](demostrable at least 6 hours after last short acting B-2 agonist use or 12 hours after last long B-2 acting agonist use).

Exclusion Criteria:

* Females of childbearing potential: pregnancy, birth control,breast-feeding
* Concurrent diseases/conditions and history of other diseases/conditions

  1. patients who have a positive history of significant clinical manifestations of allergy as a result of sensitization against tree pollen allergens, weed allergens and perennial allergens (e.g. Aspergillus spores, animal dander, house dust mite).
  2. patients with a history of food or drug related severe anaphylactoid or anaphylactic reaction(s).
* Ingredient hypersensitivity

  1. patients with known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study medication, any immunotherapy, or drugs related to Omalizumab (e.g., monoclonal antibodies, polyclonal gamma globulin).
  2. patients with hypersensitivity to the trail's asthma rescue- or escalation-medication or related drugs.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals, Basel +41 61 324 1111.
Locations (1):
- Novartis Investigator site, Nuremberg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Depigoid + Omalizumab: Depigoid administered in 4-week intervals using 0.5 ml of vial 2 (1000 DPP/mL). Omalizumab was given during the 2006 core study.
- Depigoid + Placebo: Depigoid dministered in 4-week intervals using 0.5 ml of vial 2 (1000 DPP/mL). Placebo was given during the 2006 core study
Period: Period 1 - 2007
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Started | 65 | 63
Completed | 62 | 57
Not Completed | 3 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 3
Period: Between Period 1 and Period 2
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Started | 62 | 57
Completed | 59 | 55
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Period 2 - 2008
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Started | 59 | 55
Completed | 52 | 53
Not Completed | 7 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Continuous [Mean (Standard Deviation); unit: years]
  2007 | 27.8 (9.9) | 30.4 (10.6) | 29.1 (10.3)
  2008 (N = 59/55/114) | 27.6 (9.9) | 30.1 (10.9) | 28.8 (10.5)
Age, Customized [Number; unit: participants] — 2007 Open Label (OL) extension phase
  participants
    <=18 years | 15 | 15 | 30
    Between 18 and 65 years | 50 | 48 | 98
    >=65 years | 0 | 0 | 0
Age, Customized [Number; unit: participants] — 2008 Open Label (OL) extension phase(N count for Depigoid+Omalizumab is 59 and for Depigoid+Placebo is 55)
  participants
    <= 18 years | 14 | 15 | 29
    Between 18 and 65 years | 45 | 40 | 85
    >= 65 years | 0 | 0 | 0
    Participated in 2007 but not in 2008 | 6 | 8 | 14
Sex/Gender, Customized [Number; unit: participants] — 2007 Open Label (OL) extension phase
  participants
    2007 Female | 28 | 27 | 55
    2007 Male | 37 | 36 | 73
Sex/Gender, Customized [Number; unit: participants] — 2008 Open Label (OL) extension phase(N count for Depigoid+Omalizumab is 59 and for Depigoid+Placebo is 55)
  participants
    2008 Female | 24 | 26 | 50
    2008 Male | 35 | 29 | 64
    Participated in 2007 but not in 2008 | 6 | 8 | 14
Race/Ethnicity, Customized [Number; unit: participants] — 2008 Open Label (OL) extension phase (N count for Depigoid+Omalizumab is 59 and for Depigoid+Placebo is 55)
  participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 59 | 54 | 113
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
    Participated in 2007 but not in 2008 | 6 | 8 | 14
Race/Ethnicity, Customized [Number; unit: participants] — 2007 Open Label (OL) extension phase
  participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 65 | 62 | 127
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Daily Symptom Load
Description: The daily symptom load (low=0, high=unbounded) represents the daily combined asthma and rhinoconjunctivitis symptom severity scores plus the daily asthma rescue medication score based on patient diary entries. A higher score indicates a worse patient asthma condition. Symptoms (e.g. - difficulty breathing, cough, tightness of chest, sneezing, itchy nose, red eyes, etc.) were evaluated daily by the patient using a 4-point scale (0=no symptom, 1=mild, 2=moderate, 3=severe). Point values were assigned by specific rescue medication usage. The daily scores were averaged over pollen days by site.
Time Frame: Recorded daily during the 2007 and 2008 pollen season
Population: Intent-to-Treat (ITT). The complete analysis population who consisted of all patients that received at least one dose of study drug was used for all efficacy and safety evaluations in this extension period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 1.25 (0.99) | 1.10 (0.99)
  2008 | 1.32 (1.74) | 0.97 (1.02)

2. Secondary Outcome: Asthma/Rhinoconjunctivitis Symptom Severity Score
Description: The symptom severity score was defined as the mean of the daily symptom severity scores (asthma symptoms during the day, asthma symptoms at night, rhinitis symptoms, and conjunctivitis symptoms) during the pollen season. The daily symptom severity scores were evaluated daily by the patient using a 4-point scale (0 = none (no symptom), 1 = mild, 2 = moderate, 3 = severe) and were recorded in a patient diary. The possible minimum value for the Asthma/Rhinoconjunctivitis Symptom Severity Score is 0, and the possible maximum value is 3. Higher values represent a worse outcome.
Time Frame: Recorded daily during the 2007 and 2008 pollen season
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 0.55 (0.40) | 0.55 (0.38)
  2008 | 0.54 (0.42) | 0.50 (0.37)

3. Secondary Outcome: Asthma/Rhinoconjunctivitis Rescue Medication Score
Description: Asthma/Rhinoconjunctivitis rescue medication score is a component of symptom load. Patients were advised that between visits they could take short acting β-2 agonist rescue medication as initial rescue medication for symptoms of intercurrent bronchospasm. Patients were advised that between visits they could take rescue medication (systemic antihistamines) on an as-needed basis for symptoms of grass pollen allergic rhinoconjunctivitis. The symptom load and all its components were based on the patient's entries in their diaries.
Time Frame: Recorded daily during the 2007 and 2008 pollen season
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 0.70 (0.80) | 0.55 (0.80)
  2008 | 0.78 (1.60) | 0.47 (0.97)

4. Secondary Outcome: Percentage of Participants by Global Evaluation of Treatment Effectiveness (GETE) Assessment Category Performed by the Investigator
Description: The investigator's assessment of the global evaluation of treatment effectiveness (GETE) using a five point scale, which evaluates change in asthma control/symptoms. GETE is scored as 1='excellent', 2='good', 3='moderate', 4='poor', 5='worsening' and (.)='missing').
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
percentage of participants
  2007: 1 = Excellent | 10.00 | 9.09
  2007:2 = Good | 70.00 | 54.55
  2007:3 = Moderate | 16.67 | 21.82
  2007:4 = Poor | 1.67 | 14.55
  2007:5 = Worsening | 1.67 | 0
  2007:(.) = Missing | 0 | 0
  2007:Responders (1+2) | 80 | 63.64
  2008: 1 = Excellent | 18.64 | 14.55
  2008:2 = Good | 49.15 | 30.91
  2008:3 = Moderate | 18.64 | 43.64
  2008:4 = Poor | 6.78 | 9.09
  2008:5 = Worsening | 0 | 0
  2008:(.) = Missing | 6.78 | 1.82
  2008:Responders (1+2) | 67.79 | 45.46

5. Secondary Outcome: Percentage of Participants by Global Evaluation of Treatment Effectiveness (GETE) Assessment Category Performed by the Patient
Description: The patient's assessment of the global evaluation of treatment effectiveness (GETE) using a five point scale, which evaluates change in asthma control/symptoms. GETE is scored as 1='excellent', 2='good', 3='moderate', 4='poor', 5='worsening' and (.)='missing').
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
percentage of participants
  2007: 1 = Excellent | 18.33 | 7.27
  2007: 2 = Good | 45.00 | 50.91
  2007: 3 = Moderate | 18.33 | 18.18
  2007: 4 = Poor | 10.00 | 21.82
  2007: 5 = Worsening | 1.67 | 0
  2007: (.) = Missing | 6.67 | 1.82
  2008: 1 = Excellent | 13.56 | 5.45
  2008: 2 = Good | 45.76 | 43.64
  2008: 3 = Moderate | 25.42 | 36.36
  2008: 4 = Poor | 6.78 | 9.09
  2008: 5 = Worsening | 1.69 | 1.82
  2008: (.) = Missing | 6.78 | 3.64

6. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: The Asthma Control Questionnaire (ACQ) was developed and validated for assessing asthma symptom control in patients in clinical trials as well as for individuals in clinical practice. It is a simple questionnaire consisting of seven questions assessing symptoms, airway caliber and rescue β2-agonist use. It uses a 7-point scale. The possible minimum value is 1, the possible maximum value is 7. Higher values represent worse asthma control and quality of life, respectively.
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 1.83 (0.68) | 1.97 (0.91)
  2008 | 1.82 (0.71) | 1.95 (0.80)

7. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma. It consists of 4 domains (symptoms, emotions, exposure to environmental stimuli and activity limitation). Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions (low=1, high=7). Higher values represent better quality of life.
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 6.19 (0.81) | 6.06 (0.98)
  2008 | 6.22 (0.77) | 6.21 (0.74)

8. Secondary Outcome: Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) is a 28-item disease specific questionnaire designed to measure functional impairments that are most important to patients with rhinoconjunctivitis. It consists of 7 domains (activities, sleep, common complaints, practical problems, nasal symptoms, ocular symptoms, and emotions). Patients recall their experiences during the previous week and to score each item on a 7-point scale. The overall RQLQ score is the mean response to all 28 questions (low=1, high=7). Higher values represent worse quality of life.
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007 | 2.07 (0.86) | 2.08 (0.95)
  2008 | 2.05 (0.99) | 1.98 (0.94)

9. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) and Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) - Clinical Differences to Baseline
Description: Both the AQLQ and RQLQ clinical differences were categorized as important, moderate, or meaningful improvement; no clinical change; meaningful, moderate, or important impairment. Clinically important differences in scores between any two assessments have been determined by the authors of the AQLQ and RQLQ. Changes in scores of 0.5 to 1.0 are considered clinically meaningful; 1.0 to 1.5 as moderate and > 1.5 as marked clinically important differences for any individual domain or for the overall summary score.
Time Frame: Baseline of core study and 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
participants
  2007 AQLQ: important improvement | 2 | 3
  2007 AQLQ: moderate improvement | 4 | 3
  2007 AQLQ: meaningful improvement | 8 | 4
  2007 AQLQ: no clinical change | 34 | 27
  2007 AQLQ: meaningful impairment | 5 | 9
  2007 AQLQ: moderate impairment | 2 | 4
  2007 AQLQ: important impairment | 4 | 5
  2007 AQLQ: missing | 1 | 0
  2007 RQLQ: important improvement | 4 | 3
  2007 RQLQ: moderate improvement | 4 | 3
  2007 RQLQ: meaningful improvement | 5 | 4
  2007 RQLQ: no clinical change | 27 | 25
  2007 RQLQ: meaningful impairment | 7 | 10
  2007 RQLQ: moderate impairment | 8 | 5
  2007 RQLQ: important impairment | 4 | 5
  2007 RQLQ: missing | 1 | 0
  2008 AQLQ: important improvement | 2 | 4
  2008 AQLQ: moderate improvement | 3 | 2
  2008 AQLQ: meaningful improvement | 6 | 4
  2008 AQLQ: no clinical change | 36 | 28
  2008 AQLQ: meaningful impairment | 2 | 9
  2008 AQLQ: moderate impairment | 3 | 4
  2008 AQLQ: important impairment | 4 | 3
  2008 AQLQ: missing | 3 | 1
  2008 RQLQ: important improvement | 2 | 3
  2008 RQLQ: moderate improvement | 2 | 2
  2008 RQLQ: meaningful improvement | 7 | 7
  2008 RQLQ: no clinical change | 26 | 22
  2008 RQLQ: meaningful impairment | 9 | 12
  2008 RQLQ: moderate impairment | 6 | 3
  2008 RQLQ: important impairment | 4 | 5
  2008 RQLQ: missing | 3 | 1

10. Secondary Outcome: Work Productivity and Activity Impairment
Description: The Work Productivity and Activity Impairment questionnaire measures time missed from work, impairment of work and regular activities. It consists of 6 items. The outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. The minimum value is 0 (0 %), the maximum value is 1 (100%). The recall time is 1 week. For this study WPAI-AA was used defining the specific health problem as allergic asthma, which has been validated by the instrument owner.
Time Frame: 52 Weeks (2007) and 104 Weeks (2008) after completion of core study
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
units on a scale
  2007: Work time missed due to asthma | 0.00 (0.01) | 0.01 (0.04)
  2007: Impairment while working due to asthma | 0.17 (0.20) | 0.09 (0.16)
  2007: Overall work impairment due to asthma | 0.17 (0.20) | 0.10 (0.17)
  2007: Activitiy impairment due to asthma | 0.15 (0.15) | 0.17 (0.22)
  2007Time in school activities missed due to asthma | 0.00 (0.00) | 0.01 (0.02)
  2007:Impairment in school activities due to asthma | 0.04 (0.09) | 0.11 (0.18)
  2007: Overall impairment/activities due to asthma | 0.00 (0.00) | 0.01 (0.03)
  2008: Work time missed due to asthma | 0.00 (0.01) | 0.04 (0.18)
  2008: Impairment while working due to asthma | 0.11 (0.13) | 0.10 (0.16)
  2008: Overall work impairment due to asthma | 0.11 (0.14) | 0.10 (0.16)
  2008: Activitiy impairment due to asthma | 0.16 (0.18) | 0.15 (0.19)
  2008Time in school activities missed due to asthma | 0.00 (0.00) | 0.00 (0.00)
  2008:Impairment in school activities due to asthma | 0.05 (0.06) | 0.14 (0.30)
  2008: Overall impairment/activities due to asthma | 0.00 (0.00) | 0.00 (0.00)

11. Secondary Outcome: Lung Function as Assessed by Forced Expiratory Volume in One Second (FEV1)
Description: The spirometric parameter Forced Expiratory Volume in One Second (FEV1) was measured during grass pollen season before each injection of Depigoid.
Time Frame: Assist during 2007 and 2008 pollen season
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
milliliters (mL)
  2007: FEV1 (best test) | 3886 (740) | 3661 (720)
  2008: FEV1 (best test) | 3814 (721) | 3574 (691)

12. Secondary Outcome: Lung Function as Assessed by Peak Expiratory Flow (PEF)
Description: The spirometric parameter Peak Expiratory Flow (PEF) was measured during grass pollen season before each injection of Depigoid. PEF was collected in the patient diary at seven days after visit 22, 23 and 24 as well as 35, 36 and 37. For analyzing purposes these data were averaged after the respective visits. Missing PEF-values from the patient diary were not replaced.
Time Frame: Assist during 2007 and 2008 pollen season
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: liters per minute (L/min)
Arm/Group | Depigoid + Omalizumab | Depigoid + Placebo
Number analyzed (Participants) | 60 | 55
liters per minute (L/min)
  2007: PEF (V23 or 36) | 465.6 (111.5) | 441.0 (111.8)
  2008: PEF (V23 or 36) | 463.9 (113.2) | 446.1 (116.4)

ADVERSE EVENTS:
Groups:
- Depigoid + Omalizumab 2007; Depigoid + Omalizumab 2008: Depigoid administered in 4-week intervals using 0.5 ml of vial 2 (1000 DPP/mL). Omalizumab was given during the 2006 core study.
- Depigoid + Placebo 2007; Depigoid + Placebo 2008: Depigoid dministered in 4-week intervals using 0.5 ml of vial 2 (1000 DPP/mL). Placebo was given during the 2006 core study
Arm/Group | Depigoid + Omalizumab 2007 | Depigoid + Omalizumab 2008 | Depigoid + Placebo 2007 | Depigoid + Placebo 2008
Serious Adverse Events (participants affected / at risk) | 2/65 | 5/59 | 2/63 | 1/55
Other Adverse Events (participants affected / at risk) | 36/65 | 32/59 | 34/63 | 26/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depigoid + Omalizumab 2007 (N=65) | Depigoid + Omalizumab 2008 (N=59) | Depigoid + Placebo 2007 (N=63) | Depigoid + Placebo 2008 (N=55)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depigoid + Omalizumab 2007 (N=65) | Depigoid + Omalizumab 2008 (N=59) | Depigoid + Placebo 2007 (N=63) | Depigoid + Placebo 2008 (N=55)
Conjunctivitis allergic (Eye disorders) | 2 | 0 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Injection site reaction (General disorders) | 11 | 5 | 10 | 8
Pyrexia (General disorders) | 0 | 1 | 0 | 3
Hypersensitivity (Immune system disorders) | 3 | 3 | 2 | 1
Bronchitis (Infections and infestations) | 6 | 3 | 3 | 5
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 19 | 19 | 14 | 12
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 3
Rhinitis (Infections and infestations) | 4 | 1 | 7 | 2
Sinusitis (Infections and infestations) | 3 | 6 | 2 | 4
Tonsillitis (Infections and infestations) | 0 | 3 | 4 | 2
Headache (Nervous system disorders) | 2 | 4 | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 4 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5 | 3

LIMITATIONS AND CAVEATS:
Study Start Date: February 2006 (core study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.